CLINICAL TRIAL: NCT02603679
Title: PREDIX Luminal B - Neoadjuvant Response-guided Treatment of ER Positive Tumors With High Proliferation or Low Proliferation With Metastatic Nodes. Part of a Platform of Translational Phase II Trials Based on Molecular Subtypes
Brief Title: Neoadjuvant Response-guided Treatment of Luminal B-type Tumors and Luminal A-type Tumors With Node Metastases
Acronym: PREDIX LumB
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Hatschek (Other)
Responsible Party: Sponsor-Investigator, Thomas Hatschek, Sen. Consultant, MD, PhD, Assoc. professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDIX LumB
Record Dates: First submitted 2015-11-04; First posted 2015-11-13 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Early-Stage Breast Carcinoma; Estrogen Receptor Positive Tumor
Keywords: Cyclin-Dependent Kinase Inhibitor p16
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Tamoxifen; palbociclib; Aromatase Inhibitors; Letrozole; Anastrozole; exemestane; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: Weekly Paclitaxel (Active Comparator): Patients receive weekly paclitaxel 80mg/m2, eventually dose-adjusted in relation to side effects, for a 12-week period. Thereafter, treatment is switched to endocrine treatment in combination with palbociclib. Pre- or perimenopausal women and all men are treated with tamoxifen, alternatively with an LHRH analogue in combination with an aromatase inhibitor (only women); postmenopausal women receive an aromatase inhibitor together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period, repeated twice during the second 12-week period
  Interventions: Drug: Paclitaxel
- B: Tamoxifen + Palbociclib (Experimental): Pre- or perimenopausal women and all men are treated with tamoxifen together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period, repeated twice during a 12-week period. Thereafter, treatment is switched to weekly paclitaxel 80mg/m2, eventually dose-adjusted in relation to side effects, for further 12 weeks.
  Interventions: Drug: Tamoxifen + Palbociclib
- B: Aromatase Inhibitor + Palbociclib (Experimental): Postmenopausal women receive an aromatase inhibitor together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period, repeated twice during a 12-week period. Thereafter, treatment is switched to weekly paclitaxel 80mg/m2, eventually dose-adjusted in relation to side effects, for further 12 weeks.
  Interventions: Drug: Aromatase Inhibitor + Palbociclib
- B: Goserelin + Aromatase Inhibitor + Palbociclib (Experimental): Pre- or perimenopausal women may be treated with goserelin and an aromatase inhibitor together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period, repeated twice during a 12-week period. Thereafter, treatment is switched to weekly paclitaxel 80mg/m2, eventually dose-adjusted in relation to side effects, for further 12 weeks.
  Interventions: Drug: Goserelin + Aromatase Inhibitor + Palbociclib

INTERVENTIONS:
Drug: Paclitaxel — Any brand of paclitaxel may be used, excluding nab-paclitaxel
  Arms: A: Weekly Paclitaxel
Drug: Tamoxifen + Palbociclib — Any brand of tamoxifen may be used
  Other Names: Tamoxifen; Ibrance
  Arms: B: Tamoxifen + Palbociclib
Drug: Aromatase Inhibitor + Palbociclib — Any brand of letrozole, anastrozole or exemestane may be used
  Other Names: Letrozole; Anastrozole; Exemestane; Ibrance
  Arms: B: Aromatase Inhibitor + Palbociclib
Drug: Goserelin + Aromatase Inhibitor + Palbociclib — Any brand of letrozole, anastrozole or exemestane may be used
  Other Names: Zoladex; Letrozole; Anastrozole; Exemestane; Ibrance
  Arms: B: Goserelin + Aromatase Inhibitor + Palbociclib

SUMMARY:
The purpose of this neoadjuvant trial is to evaluate efficacy and toxicity of chemotherapy using weekly paclitaxel (arm A) versus the combination of the cdk 4/6 inhibitor palbociclib and standard endocrine treatment (arm B). After 12 weeks treatment is switched crossover. During the 24-weekly treatment period, clinical and radiological evaluations are performed repeatedly. Switch between the treatment arms A and B is allowed in case of lack of response or due to toxicity. A translational subprotocol is a mandatory part of the study protocol, except for use of PET-CT evaluations. Postoperatively, patients receive three 3-weekly courses of chemotherapy with a combination of epirubicin and cyclophosphamide.

DETAILED DESCRIPTION:
Patients are randomized to either weekly treatment with paclitaxel (arm A) or endocrine treatment in combination with palbociclib (arm B) for 12 weeks. Choice of endocrine treatment is for pre- and perimenopausal women and all men tamoxifen 20 mg daily, alternatively for women in this age cohort, an LHRH analogue in combination with an aromatase inhibitor, for all postmenopausal women treatment with an aromatase inhibitor. The aromatase inhibitors to be used according to local practice are anastrozole 1 mg daily, exemestane 25 mg daily, or letrozole 2.5 mg daily. Pre- or perimenopausal women and all men are treated with tamoxifen, alternatively with an LHRH analogue in combination with an aromatase inhibitor (only women). Postmenopausal women receive an aromatase inhibitor.

After 12 weeks, patients without signs of disease progression (PD) are switched to either endocrine treatment in combination with palbociclib (arm A) or weekly treatment with paclitaxel (arm B) for 12 weeks. Postoperatively, patients receive three 3-weekly courses of chemotherapy with a combination of epirubicin and cyclophosphamide.

Before start, after 6, 12, 18 and 24 weeks of treatment, radiological assessments of tumor size are performed using mammography and ultrasound alt. MRI breast; PET-CT, confined to the breast and regional lymph nodes, before start, after 12 and 24 weeks, blood tests before start, after 1 week, 12, 18 and 24 weeks. Physical examinations are performed before start and then four-weekly after weeks 4, 8, 12, 16, 20 and 24 weeks of treatment.

In case of disease progression during ongoing study treatment, individualized management in the patient's best interest must be considered, in which case surgery is the primary option.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Female or male patients with breast cancer confirmed by histology
3. Tumor and blood samples available. Luminal B type confirmed by immunohistochemistry or, preferably, genomic profiling using Next-Generation Sequencingwith ER ≥120% and Ki67 ≥20% and not HER2 amplified, or, if aged 40 or younger and/or verified lymph node metastases, luminal A type, defined as ER and PR positive ≥20% and the proliferation marker Ki 67 <20% and not HER2 amplified. Any luminal B, Luminal A with verified lymph node metastases and/or aged 40 or younger
4. Age 18 years or older. Elderly patients in condition adequate for planned therapy
5. Primary breast cancer >20mm in diameter and/or verified regional lymph node metastases
6. Adequate bone marrow, renal, hepatic and cardiac functions and no other uncontrolled medical or psychiatric disorders
7. LVEF >55%
8. ECOG performance status 0-1
9. Primary breast cancer as defined in p. 5 plus at most 2 morphologically characterized well-defined distant metastases accessible for stereotactic radiotherapy, provided that this treatment is available

Exclusion Criteria:

1. Distant metastases, including node metastases in the contralateral thoracic region or in the mediastinum
2. Other malignancy diagnosed within the last five years, except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix
3. Patients in child-bearing age without adequate contraception
4. Pregnancy or lactation
5. Uncontrolled hypertension, heart, liver, kidney related or other medical or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiological Objective Response Rate after Completion of the First 12-week Period of Primary Medical Treatment | Start of treatment until 12 weeks of treatment
  Radiological response by use of mammography and ultrasound, alternatively MRI of the breast, if mammography/ultrasound does not allow for objective measurements of the primary tumor. Clinical measurements using calliper, if the tumor is palpable and tumor size cannot be estimated by radiological methods

SECONDARY OUTCOMES:
Pathological Objective Response Rate | From the date of surgery up to 4 weeks after surgery
  Presence/abscense of residual tumor in mm, fibrosis and other signs of response by histology
Sequencing of Chemotherapy versus Endocrine Treatment plus Palbociclib in relation to Radiological Objective Response Rate after Completion of the 24-week Period of Primary Medical Treatment | From start of treatment until termination of the preoperative treatment after 24 weeks
  Radiological response by use of mammography and ultrasound, alternatively MRI of the breast, if mammography/ultrasound does not allow for objective measurements of the primary tumor. Clinical measurements using calliper, if the tumor is palpable and tumor size cannot be estimated by radiological methods
Disease-Free Survival | From date of surgery until 10 years past surgery
  Disease-free survival includes all events related to breast cancer, and death from any cause during the follow-up period
Breast Cancer-Specific Survival | From date of surgery until 10 years past surgery
  Breast cancer-specific survival includes all events related to breast cancer and death caused by breast cancer during the follow-up period
Overall Survival | From date of surgery until 10 years past surgery
  Overall survival relates to death from any cause during the follow-up period
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From start of treatment until 28 days after termination of 24 weeks of treatment. Delayed toxicity is reported until 60 months follow-up
  Safety will be assessed using NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE) for reporting laboratory and non-laboratory toxicities
Health-Related Quality of Life | From start of study treatment until termination after 24 weeks, and then annually during 5 years of postoperative follow-up period
Frequency of Breast-Conserving Surgery | At surgery after neoadjuvant therapy
  Refers to the rate of patients who are operated with breast-conserving surgery compared with mastectomy
Characteristics of the Genome of Previously Untreated Tumors Before and After Exposition to Treatment | Before start and during treatment, at surgery, and then annually during the 60 months of postoperative follow-up period
  New Generation Sequencing (NGS) is performed on biopsies from the tumors with the aim to classify the tumors according to PAM50. Repeated analyses of tumor tissue during the treatment process will be performed to identify heterogeneity and mutations which might be responsible for resistance to study treatment. Blood samples are collected to identify tumor DNA sequences which might predict recurrence during the follow-up period. Tissue and blood samples are also analyzed in case of recurrence. The results are descriptive and expressed as clustering. Units of measure are lacking
Changes of the Proteome of Previously Untreated Tumors Before and After Exposition to Treatment | Before start, during treatment and at surgery
  Proteome analyses with the intention to identify tumor-specific pathways are performed on repeated biopsies from the tumors. The results are descriptive, defined units of measure are lacking
Quantification of Hormone Receptors Before and After Treatment | Before start, during treatment and at surgery
  Immunohistochemistry on core biopsies before start, after 10 weeks of treatment, and tumor samples from the surgical specimen. Presence of estrogen receptor (ER) and progesterone receptor (PR), described as percentage in relation to the total count of tumor cells
Quantification of Proliferation Before and After Treatment | Before start, during treatment and at surgery
  Immunohistochemistry on core biopsies before start, after 10 weeks of treatment, and tumor samples from the surgical specimen. Presence of cells indicating proliferation by use of Ki67, described as percentage in relation to the total count of tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hatschek, Assoc Prof, Study Chair — Breast-Sarcoma Unit, Dept. of Oncology, Karolinska University Hospital; Jonas Bergh, Professor, Study Director — Dept. of Oncology-Pathology, Karolinska Institutet
Locations (3):
- Sweden (3):
  - Södersjukhuset, Stockholm
  - Karolinska University Hospital, Stockholm
  - Capio S:t Göran Hospital, Stockholm